CLINICAL TRIAL: NCT00504582
Title: A Randomized Trial Evaluating the Use of Fibrin Tissue Adhesive Following Axillary Node Dissection in Patients With Melanoma
Brief Title: Fibrin Melanoma Axillary Node Study in Patients With Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS01-565; NCI-2012-01524 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Melanoma
Keywords: Axillary Node Dissection; Fibrin Sealant; Tisseel; Melanoma; Seroma
MeSH Terms: conditions — Melanoma; Seroma | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrin Sealant (Experimental): Tisseel applied externally to the dissected axillary area.
  Interventions: Drug: Fibrin Sealant
- No Fibrin Sealant (No Intervention)

INTERVENTIONS:
Drug: Fibrin Sealant — Tisseel applied externally to the dissected axillary area.
  Other Names: Tisseel
  Arms: Fibrin Sealant

SUMMARY:
Primary Objective:

* To determine whether the use of a fibrin sealant applied to axillary soft tissues following node dissection can result in earlier drain removal.

Secondary Objectives:

* To determine the postoperative morbidity rate using fibrin sealant following axillary node dissection.
* To assess patient-valuation of outcome by performing a cost-benefit analysis using a willingness-to-pay model.
* To determine if serum levels, lymphatic fluids level, or cutaneous expression of vascular endothelial growth factor-D (VEGF-D), vascular endothelial growth factor-C (VEGF-C) or their receptor, vascular endothelial growth factor receptor-3 (VEGFR-3) correlates with nodal tumor burden or development of lymphedema in patients with melanoma.

DETAILED DESCRIPTION:
Patients in this study are scheduled to have axillary node dissection as part of their surgery for treatment of their melanoma.

Within 2 weeks before entry into the study, patients will have a complete physical exam and medical history.

These patients will be randomly assigned (as in the toss of a coin) to one of two groups. Patients in one group will receive TISSEEL applied externally to the dissected axillary area. Patients in the other group will receive no fibrin sealant.

For patients who are admitted to the hospital, the surgical site will be monitored by the surgeon for evidence of wound complications in the first 24 hours after surgery. At the time of discharge from the hospital, patients will be instructed in drain care and how to measure the drainage each day until the drain is removed.

The contents of the drain will be collected from patients during the first day after surgery, during the first return follow-up visit to M.D. Anderson Cancer Center, and during drain removal (unless these latter 2 dates are the same).

Follow-up wound exams will be performed by the local primary physician or in the M.D. Anderson Melanoma Clinic between 1-4 weeks and 6 weeks after surgery. Participation will be over at the 6-week follow-up.

THIS IS AN INVESTIGATIONAL STUDY. The sealant is FDA approved, though its use in this study is experimental. About 115 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Part I - Inclusion Criteria, patients that consent to participate.
2. Patients with melanoma who have undergone axillary dissection within the last six months as part of their surgical treatment will be considered for the study.

Exclusion Criteria:

1. Part II - Exclusion Criteria, patients with known hypersensitivity to bovine proteins.
2. Patient has undergone prior radiation therapy to the operative site.
3. Patient is pregnant or lactating.
4. Patient is steroid dependent within prior 6 months.
5. Patient has used aspirin or other anti-platelet drug (excluding Celebrex) within seven days of operation.
6. Patient has pre-existing lymphedema.
7. Patient has other pre-existing medical conditions with evidence of organ dysfunction as determined by principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2002-05-15 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul F. Mansfield, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients with the diagnosis of melanoma undergoing axillary node dissection were screened for eligibility. If they met the eligibility criteria, were offered the study. The primary outcome is to determine whether the use of a fibrin sealant applied to axillary soft tissues following node dissection can result in earlier drain removal.
Pre-assignment Details: There were 121 total patients associated with this study. 92 patients were evaluable for the treatment study. 9 patients were inevaluable due to withdrew consent, surgery cancelled, patient elected to proceed with biopsy not surgery, not coming to MD Anderson, diagnosed with merkle cell carcinoma and sarcoma. There were 20 patients with melanoma who have undergone axillary dissection within prior six months as part of their surgical treatment who only completed the questionnaire.
Groups:
- Treatment Arm: Tisseel applied externally to the dissected axillary area. Intervention: Drug: Fibrin Sealant
- Control Arm: No Intervention: No Fibrin Sealant
- Questionnaire Only: Questionnaire only
Period: Overall Study
Arm/Group | Treatment Arm | Control Arm | Questionnaire Only
Started | 47 | 45 | 20
Completed | 46 | 45 | 20
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics not taken for the questionnaire only arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control Arm | Questionnaire Only | Total
Number analyzed (Participants) | 47 | 45 | 0 | 92
Age, Categorical [Count of Participants; unit: Participants] — Baseline characteristics not taken for the questionnaire only arm.
  Participants
    <=18 years | 0 | 0 |  | 0
    Between 18 and 65 years | 36 | 37 |  | 73
    >=65 years | 11 | 8 |  | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 |  | 20
  Male | 35 | 37 |  | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 |  | 2
  Not Hispanic or Latino | 46 | 44 |  | 90
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 1 |  | 1
  White | 47 | 44 |  | 91
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 45 |  | 92

OUTCOME MEASURES:

1. Primary Outcome: Drain Duration
Description: Number of days drain was in place
Time Frame: from surgery until drain removed, up to 40 days
Population: Data not collected for Questionnaire Only Arm.
Measure: Mean (Full Range); unit: days
Arm/Group | Treatment Arm | Control Arm | Questionnaire Only
Number analyzed (Participants) | 44 | 45 | 0
days | 23 [7 to 40] | 21 [5 to 36] |

2. Secondary Outcome: Number of Participants With Infection
Description: Number of participants with any signs of infection noted following surgery requiring intervention.
Time Frame: after surgery until the wound is healed, up to 30 days whichever is longer
Population: No data collected for Questionnaire Only Arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm | Questionnaire Only
Number analyzed (Participants) | 46 | 45 | 0
Participants | 12 | 8 | 0

ADVERSE EVENTS:
Time Frame: After surgery until the wound is healed or thirty days whichever is longer.
Description: No data collected for the Questionnaire Only Arm, therefore no adverse events to report for the Questionnaire Only Arm.
Arm/Group | Treatment Arm | Control Arm | Questionnaire Only
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/45 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/47 | 1/45 | 0/0
Other Adverse Events (participants affected / at risk) | 0/47 | 0/45 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=47) | Control Arm (N=45) | Questionnaire Only (N=0)
Infection (Infections and infestations) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-08-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT00504582/Prot_SAP_000.pdf